CLINICAL TRIAL: NCT05457218
Title: The Ability of Insect-derived Protein Supplements (IPC80 and Whole Buffalo Powder, Ynsect®) to Activate mTORC1 and Protein Synthesis in Muscle
Brief Title: Effect of Insect-derived Protein Supplements on Protein Synthesis and mTORC1 Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 220601
Record Dates: First submitted 2022-07-06; First posted 2022-07-13 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Effect of Food Supplement
Keywords: Protein synthesis; Protein supplement; mTORC1 activity; Insect-derived protein
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: Participants will consume a supplemental dose (0.25 g/kg body weight) of either IPC80, Whole Buffalo Powder or whey protein.
  The type of consumed supplementation will be randomized where neither the participant nor investigator will know which supplement is being consumed. Each participant will repeat the protocol three times.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A randomized double-blind crossover design with neither the subjects nor the investigators knowing who is on which treatment. The interventions will be coded using a blinded alphabetical letter code (A, B, C). A delegate researcher (independent party not further involved in the study) will randomize all interventions using a computer-generated randomization list. The delegate will hand in the code-breaker to the principal investigator in a sealed envelope. The envelope will be stored in a locked filing cabinet in the principal investigator's office, which will also be locked when unoccupied. The envelope will be opened by the principal investigator after completing the analysis of blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey protein (Experimental): This arm will be given a supplemental dose of whey protein (0.25 g/kg body weight)
  Interventions: Dietary Supplement: Whey protein
- IPC80 (Experimental): This arm will be given a supplemental dose of IPC80, an insect-derived protein source (0.25 g/kg body weight)
  Interventions: Dietary Supplement: IPC80
- Whole Buffalo Powder (Experimental): This arm will be given a supplemental dose of Whole Buffalo Powder, an insect-derived protein source (0.25 g/kg body weight)
  Interventions: Dietary Supplement: Whole Buffalo Powder

INTERVENTIONS:
Dietary Supplement: Whey protein — The participant will consume a supplemental dose of whey protein (0.25 g/kg body weight)
  Arms: Whey protein
Dietary Supplement: IPC80 — The participant will consume a supplemental dose of IPC80 (0.25 g/kg body weight)
  Arms: IPC80
Dietary Supplement: Whole Buffalo Powder — The participant will consume a supplemental dose of Whole Buffalo Powder (0.25 g/kg body weight)
  Arms: Whole Buffalo Powder

SUMMARY:
The purpose of this study is to determine the ability of insect-derived protein supplements (IPC80 and Whole Buffalo Powder Ynsect®) to activate the mTORC1 pathway and protein synthesis in muscle cells.

To achieve this aim, participants will consume a supplemental dose (0.25 g/kg body weight) of IPC80,Whole Buffalo Powder or whey protein. Blood samples will be drawn before and 15, 30, 60 and 90 minutes after the supplementation.

Protein synthesis will be assessed using stably transfected C2C12 muscle cells with a plasmid (pcDNA3 luciferase) and to determine the ability of a protein source to activate mTORC1, stably transfected C2C12 muscle cells with a plasmid (pcDNA3-TOP luciferase) where the luciferase mRNA contains a 5'TOP. 5'TOP which is specifically regulated by mTORC1 activity will be used.

DETAILED DESCRIPTION:
The purpose of this study is to determine the ability of insect-derived protein supplements (IPC80 and Whole Buffalo Powder, Ynsect®) to activate the mTORC1 pathway and protein synthesis in muscle cells.

To achieve this aim, participants will consume a supplemental dose (0.25 g/kg body weight) of IPC80, Whole Buffalo Powder or whey protein. Blood samples will be drawn before and 15, 30, 60 and 90 minutes after the supplementation.

It is expected that this project will determine whether insect-derived protein supplements (IPC80 and Whole Buffalo Powder, Ynsect®) have the ability to induce activation of the mTORC1 pathway and protein synthesis in muscle cells. Results from this study will give further insight into the usage of this novel sustainable protein source to support muscle protein synthesis after exercise.

Male and female participants between the ages of 18-30 years of age will be enrolled in the study. The study is a randomized double-blind crossover design with neither the subjects nor the investigators knowing who is on which treatment (IPC80, Whole Buffalo Powder or Whey).

I. Baseline blood draw The subjects will arrive in the laboratory following an overnight fast. The antecubital vein will be cannulated, and an initial 5 mL baseline blood sample will be collected.

II. Supplementation After baseline blood draw, subjects will be provided with a supplement, 0.25 g/kg body weight of either whey protein, IPC80 or Whole Buffalo Powder dissolved in 250ml of water.

III. Postprandial blood draws Following consumption of the supplement, the participants will remain in the laboratory for another 1.5 hours, they may bring books or electronic devices to pass the time. Four more blood samples of 5 mL each will be obtained at 15, 30, 60, and 90 minutes after supplementation, totaling five blood draws of 5mL per visit (25mL per visit), and 75 mL of blood drawn in total for each subject completing the entire study.

Blood will be collected in 5 mL serum separating tubes. All blood samples will be allowed to clot for 1hr before centrifugation at 1000 x g for 10 minutes and the serum will be frozen and kept at -30°C until processed. Treatments will be randomized to avoid an order effect and a washout period of at least 48h between trials will be used to minimize the effect of the previous treatment.

To determine protein synthesis, we have stably transfected C2C12 muscle cells with a plasmid (pcDNA3 luciferase) that we use to measure global protein synthesis. C2C12Luc cells will be plated in 24-well plates and differentiated over 4 days. Differentiated C2C12 cells will be fasted by washing with PBS and then treating them with Test Media (20% DMEM; 80% Hank's buffered salt solution (HBSS)) for 15 minutes. Fasted muscle cells will then be treated with Test Media containing 0, 2.5, 5, or 10% baseline or fed serum for 60 minutes. Cells will be collected in passive lysis buffer and firefly luciferase activity will be determined as described previously (Philp et al., 2013).

To determine the ability of a protein source to activate mTORC1 we have stably transfected C2C12 muscle cells with a plasmid (pcDNA3-TOP luciferase) where the luciferase mRNA contains a 5' terminal polypyrimidine tract (TOP). 5'TOP mRNA are specifically regulated by mTORC1 activity (Jefferies et al., 1994). As above, differentiated C2C12TOPLuc muscle cells in 24-well plates will be stimulated using the baseline or fed serum as described above. The degree of mTORC1 activation will be determined as the difference in slopes between the baseline and fed sera. The induction of mTORC1 and protein synthesis by whey and IPC80 and Whole Buffalo Powder will be compared directly within individuals and then across groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy active male or female
* Normal weight (BMI between 18 and 25 kg/m2)

Exclusion Criteria:

* Receiving any medication that may interfere with the study.
* Health or dietary restrictions that would be affected by the supplementation protocol.
* Allergy to shellfish (the chitins in the mealworm exoskeleton can activate shellfish allergies)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | Baseline (0 hour) to 15 minutes after supplementation
  To measure muscle protein synthesis, stably transfected C2C12 muscle cells with a plasmid (pcDNA3 luciferase) will be used. C2C12Luc cells will be plated in 24-well plates and differentiated over 4 days. Differentiated C2C12 cells will be fasted by washing with PBS and then treating them with Test Media (20% DMEM) for 15 minutes. Fasted muscle cells will then be treated with Test Media containing 0, 2.5, 5, or 10% baseline or fed serum (from blood samples at 15, 30, 60, and 90 minutes after supplementation) for 60 minutes. Cells will be collected in passive lysis buffer and firefly luciferase activity will be determined.
Muscle protein synthesis | Baseline (0 hour) to 30 minutes after supplementation
  To measure muscle protein synthesis, stably transfected C2C12 muscle cells with a plasmid (pcDNA3 luciferase) will be used. C2C12Luc cells will be plated in 24-well plates and differentiated over 4 days. Differentiated C2C12 cells will be fasted by washing with PBS and then treating them with Test Media (20% DMEM) for 15 minutes. Fasted muscle cells will then be treated with Test Media containing 0, 2.5, 5, or 10% baseline or fed serum (from blood samples at 15, 30, 60, and 90 minutes after supplementation) for 60 minutes. Cells will be collected in passive lysis buffer and firefly luciferase activity will be determined.
Muscle protein synthesis | Baseline (0 hour) to 60 minutes after supplementation
  To measure muscle protein synthesis, stably transfected C2C12 muscle cells with a plasmid (pcDNA3 luciferase) will be used. C2C12Luc cells will be plated in 24-well plates and differentiated over 4 days. Differentiated C2C12 cells will be fasted by washing with PBS and then treating them with Test Media (20% DMEM) for 15 minutes. Fasted muscle cells will then be treated with Test Media containing 0, 2.5, 5, or 10% baseline or fed serum (from blood samples at 15, 30, 60, and 90 minutes after supplementation) for 60 minutes. Cells will be collected in passive lysis buffer and firefly luciferase activity will be determined.
Muscle protein synthesis | Baseline (0 hour) to 90 minutes after supplementation
  To measure muscle protein synthesis, stably transfected C2C12 muscle cells with a plasmid (pcDNA3 luciferase) will be used. C2C12Luc cells will be plated in 24-well plates and differentiated over 4 days. Differentiated C2C12 cells will be fasted by washing with PBS and then treating them with Test Media (20% DMEM) for 15 minutes. Fasted muscle cells will then be treated with Test Media containing 0, 2.5, 5, or 10% baseline or fed serum (from blood samples at 15, 30, 60, and 90 minutes after supplementation) for 60 minutes. Cells will be collected in passive lysis buffer and firefly luciferase activity will be determined.

SECONDARY OUTCOMES:
mTORC1 activity | Baseline (0 hour) to 15 minutes after supplementation
  To measure the ability of a protein source (whey protein, IPC80 or Whole Buffalo Powder) to activate mTORC1, stably transfected C2C12 muscle cells with a plasmid (pcDNA3-TOP luciferase) where the luciferase mRNA contains a 5'TOP. 5'TOP mRNA , which specifically regulated by mTORC1 activity, will be used. Differentiated C2C12TOPLuc muscle cells in 24-well plates will be stimulated using the baseline or fed serum (rom blood samples at 15, 30, 60, and 90 minutes after supplementation). The degree of mTORC1 activation will be determined as the difference in slopes between the baseline and fed sera.
mTORC1 activity | Baseline (0 hour) to 30 minutes after supplementation
  To measure the ability of a protein source (whey protein, IPC80 or Whole Buffalo Powderl) to activate mTORC1, stably transfected C2C12 muscle cells with a plasmid (pcDNA3-TOP luciferase) where the luciferase mRNA contains a 5'TOP. 5'TOP mRNA , which specifically regulated by mTORC1 activity, will be used. Differentiated C2C12TOPLuc muscle cells in 24-well plates will be stimulated using the baseline or fed serum (rom blood samples at 15, 30, 60, and 90 minutes after supplementation). The degree of mTORC1 activation will be determined as the difference in slopes between the baseline and fed sera.
mTORC1 activity | Baseline (0 hour) to 60 minutes after supplementation
  To measure the ability of a protein source (whey protein, IPC80 or Whole Buffalo Powder) to activate mTORC1, stably transfected C2C12 muscle cells with a plasmid (pcDNA3-TOP luciferase) where the luciferase mRNA contains a 5'TOP. 5'TOP mRNA , which specifically regulated by mTORC1 activity, will be used. Differentiated C2C12TOPLuc muscle cells in 24-well plates will be stimulated using the baseline or fed serum (rom blood samples at 15, 30, 60, and 90 minutes after supplementation). The degree of mTORC1 activation will be determined as the difference in slopes between the baseline and fed sera.
mTORC1 activity | Baseline (0 hour) to 90 minutes after supplementation
  To measure the ability of a protein source (whey protein, IPC80 or Whole Buffalo Powder) to activate mTORC1, stably transfected C2C12 muscle cells with a plasmid (pcDNA3-TOP luciferase) where the luciferase mRNA contains a 5'TOP. 5'TOP mRNA , which specifically regulated by mTORC1 activity, will be used. Differentiated C2C12TOPLuc muscle cells in 24-well plates will be stimulated using the baseline or fed serum (rom blood samples at 15, 30, 60, and 90 minutes after supplementation). The degree of mTORC1 activation will be determined as the difference in slopes between the baseline and fed sera.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, PhD, Principal Investigator — UC Davis
Locations (1):
- Hickey Laboratory, Davis, California, United States

REFERENCES:
- [Background] Philp A, MacKenzie MG, Belew MY, Towler MC, Corstorphine A, Papalamprou A, Hardie DG, Baar K. Glycogen content regulates peroxisome proliferator activated receptor- partial differential (PPAR- partial differential) activity in rat skeletal muscle. PLoS One. 2013 Oct 17;8(10):e77200. doi: 10.1371/journal.pone.0077200. eCollection 2013. PMID 24146969
- [Background] Jefferies HB, Reinhard C, Kozma SC, Thomas G. Rapamycin selectively represses translation of the "polypyrimidine tract" mRNA family. Proc Natl Acad Sci U S A. 1994 May 10;91(10):4441-5. doi: 10.1073/pnas.91.10.4441. PMID 8183928